CLINICAL TRIAL: NCT00005878
Title: Chemoprevention for Barrett's Esophagus Trial (CBET)
Brief Title: Celecoxib to Prevent Cancer in Patients With Barrett's Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: JHOC-J9932, CDR0000067917; P30CA006973 (NIH); JHOC-J9932; JHOC-99061108; NCI-P00-0145
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Celecoxib may be effective in preventing cancer in patients with Barrett's esophagus.

PURPOSE: Randomized phase II trial to study the effectiveness of celecoxib in preventing cancer in patients who have Barrett's esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of celecoxib for regression of Barrett's dysplasia in patients with low or high-grade dysplasia of the esophagus.

OUTLINE: This is a randomized, parallel, double-blind, placebo-controlled, multicenter study. Patients are stratified according to center and grade of dysplasia at baseline (low vs high). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral celecoxib twice daily for 48-96 weeks.
* Arm II: Patients receive oral placebo as in arm I. Treatment continues in both arms in the absence of unacceptable toxicity or development of adenocarcinoma of the esophagus or cancer at other sites.

Patients are followed at 12 weeks.

PROJECTED ACCRUAL: A total of 200 patients (100 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Barrett's dysplasia with specific information on the location (level) of the highest grade of dysplasia based on biopsy from baseline endoscopy

  * Short segment Barrett's esophagus must be sufficient area to allow for biopsy without complete resection
* No presence of reflux esophagitis grades 2-4
* No history of confirmed invasive carcinoma of the esophagus
* No diagnosis of esophageal, gastric, pyloric channel, or duodenal ulceration of 1 cm or more in diameter within the past 30 days

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 9 g/dL
* Platelet count greater than 125,000/mm^3
* WBC greater than 3,000/mm^3
* No significant bleeding disorder
* No other abnormal hematopoietic laboratory test result that would preclude study

Hepatic:

* PT/PTT no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT less than 1.5 times ULN
* Alkaline phosphatase less than 1.5 times ULN
* No chronic or acute hepatic disorder
* No abnormal hepatic laboratory test result that would preclude study

Renal:

* Creatinine no greater than 1.5 times ULN
* No chronic or acute renal disorder
* No other abnormal renal laboratory test result that would preclude study

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior or concurrent active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
* No other prior or concurrent curatively treated malignancy with a survival prognosis of less than 5 years
* No hypersensitivity or adverse reaction to COX-2 inhibitors (e.g., celecoxib), sulfonamides, salicylates, or NSAIDs
* No other significant medical, psychological, or psychosocial condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 6 months since prior regular (at least 2 weeks duration) oral or intravenous corticosteroids
* At least 6 months since prior regular (at least 4 weeks duration) inhaled corticosteroids
* No concurrent regular oral or intravenous corticosteroids
* No concurrent regular inhaled corticosteroids
* Concurrent corticosteroid nasal spray allowed

Radiotherapy:

* At least 12 weeks since prior radiotherapy to the chest or upper abdomen

Surgery:

* At least 3 months since prior surgery to the esophagus or stomach except hiatal hernia repair, fundoplication, vagotomy, or pyloroplasty
* No prior complete mucosal resection using any technique
* No concurrent resection of high-grade nodule

Other:

* At least 30 days since prior chronic (at least 3 times a week for greater than 2 weeks) aspirin or other nonsteroidal antiinflammatory drugs (NSAIDs) (i.e., greater than 100 mg/day)
* No prior complete mucosal ablation using any technique
* No prior treatment on this study
* At least 30 days since prior investigational medication including shingles vaccine
* No concurrent chronic NSAIDs or COX-2 inhibitors except low-dose aspirin (i.e., no greater than 100 mg/day)
* No concurrent anticoagulants (e.g., heparin or warfarin)
* No other concurrent investigational medication

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (8):
- United States (8):
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Portland, Portland, Oregon

REFERENCES:
- [Result] Heath EI, Canto MI, Piantadosi S, Montgomery E, Weinstein WM, Herman JG, Dannenberg AJ, Yang VW, Shar AO, Hawk E, Forastiere AA; Chemoprevention for Barrett's Esophagus Trial Research Group. Secondary chemoprevention of Barrett's esophagus with celecoxib: results of a randomized trial. J Natl Cancer Inst. 2007 Apr 4;99(7):545-57. doi: 10.1093/jnci/djk112. PMID 17405999